CLINICAL TRIAL: NCT00552110
Title: Efficacy and Safety of Concurrent Administration of Mometasone Furoate Nasal Spray (MFNS) and Oxymetazoline Nasal Spray Administered Once Daily (QD) vs. Oxymetazoline Twice Daily (BID), Mometasone Furoate QD, and Placebo in the Treatment of Subjects With Seasonal Allergic Rhinitis
Brief Title: Study of Mometasone Furoate Nasal Spray and Oxymetazoline Nasal Spray Given Together Once A Day To Treat Seasonal Allergic Rhinitis (P04500)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P04500
Record Dates: First submitted 2007-10-30; First posted 2007-11-01 (Estimated); Results first posted 2009-07-08 (Estimated); Last update posted 2024-05-14 (Actual); Status verified 2022-02

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Combination1 (Experimental): Mometasone Furoate nasal spray (MFNS) with oxymetazoline nasal spray (OXY) 1 spray once daily
  Interventions: Drug: OXY combination: mometasone furoate nasal spray (MFNS) and oxymetazoline nasal spray (OXY)
- Combination3 (Experimental): MFNS with OXY 3 sprays once daily
  Interventions: Drug: OXY combination: mometasone furoate nasal spray (MFNS) and oxymetazoline nasal spray (OXY)
- Mometasone (Active Comparator): MFNS once daily
  Interventions: Drug: mometasone furoate nasal spray (MFNS) once daily
- Oxymetazoline (Active Comparator): OXY twice daily
  Interventions: Drug: oxymetazoline nasal spray (OXY) twice daily
- Placebo (Placebo Comparator): Placebo nasal spray
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OXY combination: mometasone furoate nasal spray (MFNS) and oxymetazoline nasal spray (OXY) — MFNS 2 sprays per nostril with OXY 1 spray per nostril once daily x 2 weeks. Matching placebo to MFNS given every evening (PM).
  Other Names: MFNS + OXY combination
  Arms: Combination1
Drug: OXY combination: mometasone furoate nasal spray (MFNS) and oxymetazoline nasal spray (OXY) — MFNS 2 sprays per nostril with OXY 3 sprays per nostril once daily x 2 weeks. Matching placebo to MFNS given every evening.
  Other Names: MFNS + OXY combination assessing a different dose (ie, number of sprays) from that used in Group 1
  Arms: Combination3
Drug: mometasone furoate nasal spray (MFNS) once daily — MFNS 2 sprays per nostril once daily x 2 weeks. Matching placebo to MFNS given every morning (AM) and every evening.
  Other Names: MFNS QD
  Arms: Mometasone
Drug: oxymetazoline nasal spray (OXY) twice daily — OXY 2 sprays per nostril twice daily x 2 weeks. Matching placebo to MFNS given every morning.
  Other Names: OXY BID
  Arms: Oxymetazoline
Drug: Placebo — Matching placebo to MFNS given every morning and every evening x 2 weeks.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the efficacy of the combination of mometasone furoate nasal spray (MFNS) and oxymetazoline nasal spray (OXY) given together once a day in treating subjects with seasonal allergic rhinitis (SAR) in relieving symptoms including nasal congestion. The secondary objectives of this study are to evaluate the potential of the combination to produce tachyphylaxis and/or rebound congestion, and to evaluate the safety of the combination.

ELIGIBILITY:
Inclusion Criteria:

* Must be 12 years of age or older, of either sex, and of any race.
* Must have at least a 2-year documented history of SAR which exacerbates during the time period over which the subject will be participating.
* Must have a documented (within the past 12 months) positive skin-prick test response to an appropriate seasonal allergen appropriate to the geographical vicinity in which the study is being carried out and over the period of time the subject is participating.
* Must be clinically symptomatic at the Screening and Baseline Visits.
* Must be in general good health as confirmed by routine clinical and laboratory testing and electrocardiogram results.
* Must be free of any clinically significant disease, other than SAR, which would interfere with the study evaluations.
* Must be willing to give written informed consent and must be able to adhere to dosing and visit schedules and study requirements.
* Female subjects of child-bearing potential must have a negative serum pregnancy test at screening. Nonsterile and premenopausal female subjects must be using a medically acceptable method of birth control prior to screening and during the entire study.
* Must have the ability to transmit electronic diary data on a regular basis.

Exclusion Criteria:

* A subject with a history of anaphylaxis and/or other severe local reaction(s) to skin testing.
* A subject with asthma who requires chronic use of inhaled or systemic corticosteroids.
* A subject with current or history of frequent, clinically significant sinusitis or chronic purulent postnasal drip.
* A subject with rhinitis medicamentosa.
* A subject with glaucoma and/or increased intraocular pressure.
* A subject who has nasal structural abnormalities, including large nasal polyps and marked septal deviations, which significantly interfere with nasal air flow.
* A subject who, in the opinion of the investigator, is dependent on nasal, oral, or ocular decongestants, nasal topical antihistamines, or nasal steroids.
* A pregnant or nursing female.
* A subject with current evidence of clinically significant hematopoietic, cardiovascular, hepatic, renal, neurologic, psychiatric, pulmonary, autoimmune disease, or other disease that precludes the subject's participation in the study. Particular attention should be given to exclude subjects with conditions that would currently interfere with the absorption, distribution, metabolism, or excretion of the study drug or interfere with the subject's ability to complete or reliably complete the diaries.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 707 (Actual)
Dates: Start 2007-07; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariel A Teper, MD, Study Director — Schering-Plough

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Meltzer EO, Bernstein DI, Prenner BM, Berger WE, Shekar T, Teper AA. Mometasone furoate nasal spray plus oxymetazoline nasal spray: short-term efficacy and safety in seasonal allergic rhinitis. Am J Rhinol Allergy. 2013 Mar-Apr;27(2):102-8. doi: 10.2500/ajra.2013.27.3864. PMID 23562197

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Combination1 | Combination3 | Mometasone | Oxymetazoline | Placebo
Started | 146 (One subject was excluded from the intent to treat population because there was no record of dosing.) | 139 | 139 | 141 (One subject was excluded from the intent to treat population because there was no record of dosing.) | 142
Completed | 142 | 134 | 137 | 133 | 133
Not Completed | 4 | 5 | 2 | 8 | 9
Not completed — Serious or Life-Threatening AE | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 1 | 4
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 3 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 1
Not completed — Failed to Comply With Study Requirements | 1 | 1 | 1 | 0 | 1
Not completed — Withdrawn per Sponsor | 0 | 1 | 0 | 0 | 1
Not completed — Use of Prohibited Medication | 1 | 1 | 0 | 0 | 0
Not completed — Delay of Study due to Relabeling | 0 | 0 | 0 | 1 | 0
Not completed — Increased Blood Pressure at Visit 2 | 0 | 0 | 0 | 1 | 0
Not completed — Nonserious Adverse Event (AE) | 1 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combination1 | Combination3 | Mometasone | Oxymetazoline | Placebo | Total
Number analyzed (Participants) | 145 | 139 | 139 | 140 | 142 | 705
Age, Categorical [Count of Participants; unit: Participants] — Intention to treat population: all randomized subjects who had taken at least one dose of study drug
  Participants
    <=18 years | 8 | 12 | 5 | 5 | 12 | 42
    Between 18 and 65 years | 135 | 124 | 132 | 131 | 127 | 649
    >=65 years | 2 | 3 | 2 | 4 | 3 | 14
Sex: Female, Male [Count of Participants; unit: Participants] — Intention to treat population: all randomized subjects who had taken at least one dose of study drug
  Participants
    Female | 93 | 93 | 101 | 95 | 89 | 471
    Male | 52 | 46 | 38 | 45 | 53 | 234

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in AM/PM Instantaneous Total Nasal Symptom Score (NOW TNSS) Averaged Over Days 1 to 15
Description: Subjects scored severity of rhinorrhea, nasal congestion/stuffiness, nasal itching, and sneezing at the time of evaluation (NOW) using an ordinal scale from 0 = none to 3 = severe. Evaluations were performed daily in the morning (AM) and evening (PM). For each evaluation, individual symptom scores were summed to a TNSS, which was then averaged for a single score across the 15 day treatment period.
Time Frame: 15 days of treatment
Population: Intention to treat (ITT): all randomized subjects who had taken at least one dose of study drug
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Combination1 | Combination3 | Mometasone | Oxymetazoline | Placebo
Number analyzed (Participants) | 145 | 138 | 139 | 139 | 140
units on a scale | -3.29 (0.209) | -3.36 (0.216) | -2.97 (0.213) | -2.44 (0.215) | -1.90 (0.209)
Statistical Analysis 1: Comparison: Combination1 vs Oxymetazoline; Null hypothesis: the concurrent administration of MFNS and OXY once daily has the same mean change from baseline in AM/PM NOW TNSS as that of OXY twice daily. Power calculation: The target randomization of 875 subjects (175 subjects per treatment arm) was needed to detect a treatment difference of 0.8 point or more in change from baseline in AM/PM NOW TNSS, with a two-sided alpha of 0.05 and 90% power, assuming a pooled standard deviation of 2.3 points; Test type: Superiority or Other; p = 0.002, ANCOVA — Multiplicity for multiple treatment comparisons was not adjusted; Analysis of Covariance (ANCOVA); classification variables: treatment, center, dosing sequence (stratification variable); covariate: baseline score
Statistical Analysis 2: Comparison: Combination3 vs Oxymetazoline; Null hypothesis: the concurrent administration of MFNS and OXY once daily has the same mean change from baseline in AM/PM NOW TNSS as that of OXY twice daily; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 3: Comparison: Mometasone vs Placebo; Null hypothesis: the administration of MFNS once daily has the same mean change from baseline in AM/PM NOW TNSS as that of placebo; Test type: Superiority or Other; p < 0.001, ANCOVA

2. Primary Outcome: Standardized Area Under the Curve From 0 to 4 Hours [AUC(0-4 hr)] of the Change From Baseline to Hour 4 on Day 1 in Nasal Congestion Score
Description: Subjects scored nasal congestion/stuffiness using an ordinal scale from 0 = none to 3 = severe. Baseline was the average of the scores assessed every 15 minutes for 1 hour prior to dosing on Day 1. After dosing on Day 1, congestion was scored every 15 minutes for the 1st hour and every 30 minutes for the next 3 hours. Area under the curve (AUC) was calculated using the trapezoid rule, then standardization achieved by dividing the calculation by 4 hours. Treatment comparisons were examined using the standardized AUC(0-4 hr) of the change from baseline to hour 4 on Day 1.
Time Frame: from baseline to hour 4 on Day 1
Population: Intention to treat: all randomized subjects who had taken at least one dose of study drug
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Combination1 | Combination3 | Mometasone | Oxymetazoline | Placebo
Number analyzed (Participants) | 144 | 138 | 139 | 139 | 140
units on a scale | -0.80 (0.056) | -0.92 (0.057) | -0.63 (0.057) | -1.06 (0.057) | -0.57 (0.056)
Statistical Analysis 1: Comparison: Combination1 vs Mometasone; Null hypothesis: the concurrent administration of MFNS and OXY once daily has the same standardized AUC(0-4 hr) of the change from baseline in nasal congestion score as that of MFNS once daily; Test type: Superiority or Other; p = 0.021, ANCOVA — Multiplicity for multiple treatment comparisons was not adjusted; ANCOVA; classification variables: treatment, center, dosing sequence (stratification variable); covariate: baseline score
Statistical Analysis 2: Comparison: Combination3 vs Mometasone; Null hypothesis: the concurrent administration of MFNS and OXY once daily has the same standardized AUC (0-4hr) of the change from baseline in nasal congestion score as that of MFNS once daily; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 3: Comparison: Oxymetazoline vs Placebo; Null hypothesis: the administration of OXY twice daily has the same standardized AUC(0-4 hr) of the change from baseline in nasal congestion score as that of placebo; Test type: Superiority or Other; p < 0.001, ANCOVA

ADVERSE EVENTS:
Arm/Group | Combination1 | Combination3 | Mometasone | Oxymetazoline | Placebo
Serious Adverse Events (participants affected / at risk) | 0/145 | 0/139 | 1/139 | 0/140 | 1/142
Other Adverse Events (participants affected / at risk) | 7/145 | 5/139 | 10/139 | 7/140 | 8/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination1 (N=145) | Combination3 (N=139) | Mometasone (N=139) | Oxymetazoline (N=140) | Placebo (N=142)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination1 (N=145) | Combination3 (N=139) | Mometasone (N=139) | Oxymetazoline (N=140) | Placebo (N=142)
Headache (Nervous system disorders) | 7 (9) | 5 (5) | 10 (11) | 7 (8) | 8 (8)

LIMITATIONS AND CAVEATS:
Subject symptom data were not collected during the post-treatment period. Thus, daily diary data for rebound congestion was not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less